CLINICAL TRIAL: NCT00917605
Title: Robot-Assisted Upper Limb Rehabilitation in Stroke
Brief Title: Robot-Assisted Therapy in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200903080R
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-03

CONDITIONS: Cerebrovascular Accidents; Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Other: Robot-assisted therapy — Patients will receive an intervention for 20 training sessions (1.5 hours/day, 5 days/week for 4 consecutive weeks). The Robot-assisted arm trainer, Bi-Manu-Track (Reha-Stim Co., Berlin, Germany), will be used in this project. The Bi-Manu-Track enables the symmetrical practice of 2 movement patterns: forearm pronation-supination and wrist flexion-extension (Hesse et al., 2003; Hesse et al., 2005). Each movement has three computer-controlled modes: (1) passive-passive, with both arms being moved by the machine with speed and range of motion individually adjustable; (2) active-passive, with the nonaffected arm driving the affected arm in a mirror-like fashion; and (3) active-active, with both arms actively moving against resistance. Mode 3 is an active mode as in 2, but the paretic arm had to overcome an individually set, initially isometric resistance to allow the bilateral movement. The speed of movement, the amount of resistance, and the range of movement can be adjusted individually.

SUMMARY:
This project consists of two parts: Robotic Rehabilitation Trials, and Study of Outcome Predictors and Clinimetric Attributes. In the first part of study, the investigators aim to (1) investigate the treatment effects of robot-assisted therapy (RAT) in patients with stroke on various outcomes, (2) test the dose-response relations by using two different intensities (higher versus lower intensity RAT), and (3) investigate the effects of the training intensity on a biomarker of oxidative stress. Treatment outcomes will encompass the spectrum of functioning including motor ability, motor control strategies, basic/extended daily functions, mobility, community reintegration, quality of life, and biomarker (8-OHdG). In the second part of study, the purposes are to define the appropriate populations for RAT and to examine the clinimetric properties of clinical measures relevant for use in robotic rehabilitation research. the investigators will identify the clinical predictors that will potentially influence the functional outcomes after interventions. Finally, the investigators will examine and compare the clinimetric properties (e.g., validity and responsiveness) of the clinical measures of rehabilitation outcome to inform selection of test instruments that may detect clinically meaningful change after rehabilitation therapy.

ELIGIBILITY:
Inclusion Criteria:

1. 3 to 24 months onset from a first-ever unilateral stroke
2. an initial UL subsection of the Fugl-Meyer Assessment score of 18 to 56 indicating moderate to severe and moderate UL movement impairment
3. no excessive spasticity in any of the joints of the affected UL (shoulder, elbow, wrist, fingers)
4. be able to follow study instructions and perform study tasks
5. without upper limb fracture within 3 months
6. lack of participation in any experimental rehabilitation or drug studies during the study period
7. willing to provide written informed consent

Exclusion Criteria:

1. subjects exhibiting physician-determined major medical problems or poor physical conditions that would interfere with participation
2. subjects with excessive pain in any joint that might limit participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment | before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Keh-chung Lin, ScD, Principal Investigator — National Taiwan University Hospltal
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Wu CY, Yang CL, Chen MD, Lin KC, Wu LL. Unilateral versus bilateral robot-assisted rehabilitation on arm-trunk control and functions post stroke: a randomized controlled trial. J Neuroeng Rehabil. 2013 Apr 12;10:35. doi: 10.1186/1743-0003-10-35. PMID 23587106
- [Derived] Chuang LL, Lin KC, Wu CY, Chang CW, Chen HC, Yin HP, Wang L. Relative and absolute reliabilities of the myotonometric measurements of hemiparetic arms in patients with stroke. Arch Phys Med Rehabil. 2013 Mar;94(3):459-66. doi: 10.1016/j.apmr.2012.08.212. Epub 2012 Sep 4. PMID 22960277
- [Derived] Hsieh YW, Wu CY, Lin KC, Yao G, Wu KY, Chang YJ. Dose-response relationship of robot-assisted stroke motor rehabilitation: the impact of initial motor status. Stroke. 2012 Oct;43(10):2729-34. doi: 10.1161/STROKEAHA.112.658807. Epub 2012 Aug 14. PMID 22895994
- [Derived] Chuang LL, Wu CY, Lin KC. Reliability, validity, and responsiveness of myotonometric measurement of muscle tone, elasticity, and stiffness in patients with stroke. Arch Phys Med Rehabil. 2012 Mar;93(3):532-40. doi: 10.1016/j.apmr.2011.09.014. Epub 2012 Jan 4. PMID 22222143